CLINICAL TRIAL: NCT06605352
Title: Clinical Impact of Rapid Molecular Testing for Pathogens in Patients With Severe Acute Respiratory Illness : A Pragmatic Trial
Acronym: CIRT-RMT-SARI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Clinical Trial Center (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201908092RIND, 2024-09-008B
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Community-Acquired Pneumonia (CAP); Pneumonia
Keywords: Community-acquired pneumonia (CAP); multiplex PCR; emergency department (ED); Pneumonia; Procalcitonin(PCT); antimicrobial resistance
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Emergencies

STUDY DESIGN:
Intervention Model Description: The BIOFIRE®FILMARRAY® Pneumonia Panel is the only FDA approved mPCR test that can test 18bacteria (11 Gram negative, 4 Gram positive and 3 atypical), 7 antibiotic resistance markers, and 9 viruses in one test within 45
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pneumonia Panel (Experimental): The BIOFIRE®FILMARRAY® Pneumonia Panel is the only FDA approved mPCR test that can test 18bacteria (11 Gram negative, 4 Gram positive and 3 atypical), 7 antibiotic resistance markers, and 9 viruses in one test within 45 minutes.
  Using rapid diagnostic test to improve the proportion of antibiotics change, including escalation, de-escalation, discontinuation, or addition of antimicrobial medications in 24 hours within sample collection.
  Interventions: Diagnostic Test: The BIOFIRE®FILMARRAY® Pneumonia Panel
- Control group (No Intervention): Using current methods (empirical antibiotics) to treat patents with suspected bacterial infections.

INTERVENTIONS:
Diagnostic Test: The BIOFIRE®FILMARRAY® Pneumonia Panel — The BIOFIRE®FILMARRAY® Pneumonia Panel is the only FDA approved mPCR test that can test 18bacteria (11 Gram negative, 4 Gram positive and 3 atypical), 7 antibiotic resistance markers, and 9 viruses in one test within 45 minutes.
  Using rapid diagnostic test to improve the proportion of antibiotics change, including escalation, de-escalation, discontinuation, or addition of antimicrobial medications in 24 hours within sample collection.
  Arms: Pneumonia Panel

SUMMARY:
Community-acquired pneumonia (CAP) is among the most common reasons for emergency department (ED) visits. A clear understanding of the likely pathogens is essential for the rapid institution of adequate antimicrobial therapy. Due to the indistinguishable clinical symptoms between viral and bacterial pathogens, patients with viral respiratory infection are usually under-evaluated while unnecessary antibacterial agents are more likely to be administered. With the development of highly sensitive end-to-end point-of-care (POC) multiplex PCR system, rapid diagnosis of respiratory pathogens for CAP in the ED becomes possible. Our previous NTUH-VGH cooperative research project demonstrated POC respiratory viral testing' in conjunction with procalcitonin test can reduce the length of hospital stay and antibiotic consumption. However, viral testing alone cannot guide precision antimicrobial treatment. A complete pneumonia pathogen testing panel should include bacteria, virus, atypical pathogens, and resistant genes. In addition, such test need to be completed within about time at a reasonable cost. The difficult missing has been recently achieved. The BIOFIRE®FILMARRAY® Pneumonia Panel is the only FDA approved mPCR test that can test 18 bacteria (11 Gram negative, 4 Gram positive and 3 atypical), 7 antibiotic resistance markers, and 9 viruses in one test within 45 minutes. Currently, the world is eagerly to learn how this new diagnostic technology can transform the clinical management of pneumonia. With this in mind, the aim of this study is to evaluate the impact of POC pneumonia pathognome wide testing on the antimicrobial use and outcome of patients. We will perform an open label pragmatic parallel comparison between patients with/without the test. The results will inform the pneumonia guideline. Subsequent health economic analysis based on this study will be important to the reimbursement policy of the health insurance of Taiwan.

DETAILED DESCRIPTION:
Community-acquired pneumonia is among the most common reasons for emergency department (ED) visits and can be caused by both viral and bacterial pathogens. A clear understanding of the likely pathogens is essential for the rapid institution of adequate antiviral or antibiotic therapy. Due to the indistinguishable clinical symptoms between viral and bacterial pathogens, patients with viral respiratory infection are usually undervalued while unnecessary antibacterial agents are more likely to be administered. The principal bacterial causes of CAP are well described, with Streptococcus pneumoniae being the most important pathogen in all age groups. Recent studies and our previous work showed viral associated CAP can be responsible for 20 to 30% of CAP. Therefore, laboratory tests providing accurate and timely determination of the infectious agents associated with CAP are important. A broad array of tests is available to detect viral respiratory agents. Rapid antigen tests are available for influenza A and B, and respiratory syncytial virus (RSV), but these tests have low sensitivity and specificity.

Molecular diagnostic tests using the polymerase chain reaction (PCR) method to detect RNA or DNA of the infectious agents have improved the ability to detect both viral and bacterial pathogens in clinical samples, but are technically challenging and time consuming. The advent of sensitive point-of-care (POC) molecular detection methods has made rapid diagnosis of respiratory virus infections possible. A POC systems that automates the real-time PCR process and integrates sample preparation, amplification, detection, and analysis into one complete process has been developed and approved by the FDA. Initial studies demonstrated that such POC multiplex PCR systems' identified previously under-evaluated viral or atypical infections in ED dyspneic patients. Despite the availability of highly accurate viral testing results, discontinuation of de-escalation of antibiotics still raises concerns because polymicrobial infections involving bacterial and viral pathogens is common in the older adults. An ideal pathogen diagnostic tool for CAP that can guide precise prescription of antibiotics should therefore include the following three features: first, including a wide array of both common viral and bacterial pathogens for CAP, second, including common drug resistance genes for bacterial pathogens, and lastly, easy operation with quick turnaround time and high accuracy.

Such diagnostic tool has recently been developed. The BIOFIRE® FILMARRAY® Pneumonia Panel plus tests for 18 bacteria (11 Gram negative, 4 Gram positive and 3 atypical), 7 antibiotic resistance markers, and 9 viruses that cause pneumonia and other lower respiratory tract infections. The target bacteria included Acinetobacter calcoaceticus-baumannii complex, Enterobacter cloacae, Escherichia coli, Haemophilus influenzae, Klebsiella aerogenes, Klebsiella oxytoca, Klebsiella pneumoniae group, Moraxella catarrhalis, Proteus spp., Pseudomonas aeruginosa, Serratia marcescens, Staphylococcus aureus, Streptococcus agalactiae, Streptococcus pneumoniae, Streptococcus pyogenes. Seven antibiotics genes include ESBL (CTX-M), Carbapenemases (KPC, NDM, Oxa48-like, VIM, IMP, Methicillin Resistance (mecA/mecC and MREJ). The atypical pathogens include Legionella pneumophila, Mycoplasma pneumoniae, and Chlamydia pneumoniae. The virus included Influenza A, Influenza B, Adenovirus, Coronavirus, Parainfluenza virus, Respiratory Syncytial virus, Human Rhinovirus/Enterovirus, Human Metapneumovirus, and even Middle East Respiratory Syndrome Coronavirus (MERS-CoV). The Filmarray system is a US FDA system that integrates sample preparation, nucleic acid extraction and purification, amplification, detection and analysis into one simple system that requires just 2 minutes of hands-on time, with a total run time of about one hour. Currently, the overall sensitivity and specificity for bronchoalveolar (BAL)-like samples of 96,2% and 98.3%, respectively, and for sputum samples a sensitivity and specificity of 96.3% and 97.2%, respectively.

In this study, we aim to assess the impact of implementation of POC molecular testing for pneumonia pathogens in conjunction with procalcitonin tests on elderly patients presenting to the ED with severe acute respiratory illness. We will conduct a prospective cohort study in the EDs of two urban medical centers. Clinical impact will be evaluated through the comparison between the experimental cohort with a randomly selected control cohort in a parallel fashion. In addition to POC molecular test, we will also test procalcitonin on these patients. With a highly sensitive POC molecular test, it is likely the detection of colonized pathogens will greatly increase. PCT is a precursor of calcitonin that is constitutively secreted by C cells of the thyroid gland and K cells of the lung. In healthy individuals, PCT is normally undetectable (below 0.01 ng/mL). When stimulated by endotoxin, PCT is rapidly produced by parenchymal tissue throughout the body. Unlike C-reactive protein, PCT does not respond to sterile inflammation or viral infection. Multiple randomized controlled trials have demonstrated that procalcitonin levels of under 0.25 µg/L can guide the decision to withhold antibiotics or stop therapy early. In addition, a procalcitonin levels of under 0.1 µg/L can indicate colonization. We hypothesize the new diagnostic approach would better guide the antibiotic treatment and ultimately improve patient's outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the ED
2. Age ≥18 years old
3. Diagnosis of SARI -modified from the World Health Organization definition:

   * history of fever or measured fever of ≥ 38 C° and cough
   * with onset within the last 10 days.
   * requires hospitalization.
   * with SpO2 on presentation less than 95% or respiratory rate more than 20 per minute, or requirement of intubation and mechanical ventilation.

Exclusion Criteria:

1. Patients receiving palliative care
2. Patients who declined sample collection
3. Patients fail to provide written informed consent.
4. Patients highly suspected or diagnosed pulmonary non-infectious disease (tumor, immune disease, etc) without evidence of infection.
5. Patients diagnosed with COVID-19 within last 3 months.
6. HIV-infected patients.
7. Off work hour collected samples will be excluded from the study.
8. Patients who died or being transitioned to comfort care within 48 hours of enrollment.

Study Population Description Inclusion criteria will be 1) ED patients age 18 or older; 2) presenting to the emergency department with acute severe respiratory illness. We define a case of severe acute respiratory illness (SARI) according to a previously suggested WHO case definition for all adults in whom onset of illness occurred within 7 days of admission. We defined SARI in adult as physician-diagnosed lower respiratory tract infection (LRTI) with SpO2 on presentation less than 95% or respiratory rate more than 20 per minute, or requirement of intubation and mechanical ventilation.

Sampling Method: random sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of antibiotics change | 2 years
  The proportion of antibiotics change, including escalation, de-escalation, discontinuation, or addition of antimicrobial medications in 24 hours within sample collection.

SECONDARY OUTCOMES:
Patients Prognosis | 2 years
  The proportion of patients re-admitted in 30 days, the average length of hospital stay, 30-day all-cause mortality, duration of intravenous antibiotics, duration of mechanical ventilator.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SH, Ruan SY, Pan SC, Lee TF, Chien JY, Hsueh PR. Performance of a multiplex PCR pneumonia panel for the identification of respiratory pathogens and the main determinants of resistance from the lower respiratory tract specimens of adult patients in intensive care units. J Microbiol Immunol Infect. 2019 Dec;52(6):920-928. doi: 10.1016/j.jmii.2019.10.009. Epub 2019 Nov 23. PMID 31806539
- [Background] Murphy CN, Fowler R, Balada-Llasat JM, Carroll A, Stone H, Akerele O, Buchan B, Windham S, Hopp A, Ronen S, Relich RF, Buckner R, Warren DA, Humphries R, Campeau S, Huse H, Chandrasekaran S, Leber A, Everhart K, Harrington A, Kwong C, Bonwit A, Dien Bard J, Naccache S, Zimmerman C, Jones B, Rindlisbacher C, Buccambuso M, Clark A, Rogatcheva M, Graue C, Bourzac KM. Multicenter Evaluation of the BioFire FilmArray Pneumonia/Pneumonia Plus Panel for Detection and Quantification of Agents of Lower Respiratory Tract Infection. J Clin Microbiol. 2020 Jun 24;58(7):e00128-20. doi: 10.1128/JCM.00128-20. Print 2020 Jun 24. PMID 32350043
- [Background] Kosai K, Akamatsu N, Ota K, Mitsumoto-Kaseida F, Sakamoto K, Hasegawa H, Izumikawa K, Mukae H, Yanagihara K. BioFire FilmArray Pneumonia Panel enhances detection of pathogens and antimicrobial resistance in lower respiratory tract specimens. Ann Clin Microbiol Antimicrob. 2022 Jun 4;21(1):24. doi: 10.1186/s12941-022-00512-8. PMID 35659683
- [Background] Buchan BW, Windham S, Balada-Llasat JM, Leber A, Harrington A, Relich R, Murphy C, Dien Bard J, Naccache S, Ronen S, Hopp A, Mahmutoglu D, Faron ML, Ledeboer NA, Carroll A, Stone H, Akerele O, Everhart K, Bonwit A, Kwong C, Buckner R, Warren D, Fowler R, Chandrasekaran S, Huse H, Campeau S, Humphries R, Graue C, Huang A. Practical Comparison of the BioFire FilmArray Pneumonia Panel to Routine Diagnostic Methods and Potential Impact on Antimicrobial Stewardship in Adult Hospitalized Patients with Lower Respiratory Tract Infections. J Clin Microbiol. 2020 Jun 24;58(7):e00135-20. doi: 10.1128/JCM.00135-20. Print 2020 Jun 24. PMID 32350045
- [Background] Jitmuang A, Puttinad S, Hemvimol S, Pansasiri S, Horthongkham N. A multiplex pneumonia panel for diagnosis of hospital-acquired and ventilator-associated pneumonia in the era of emerging antimicrobial resistance. Front Cell Infect Microbiol. 2022 Oct 12;12:977320. doi: 10.3389/fcimb.2022.977320. eCollection 2022. PMID 36310855
- See also: BioFire pneumonia panel website — https://www.biomerieux.com/us/en/our-offer/clinical-products/biofire-pneumonia-panel.html